CLINICAL TRIAL: NCT01229501
Title: Fat Biology, Sleep Disorders, and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, PI, Mayo Clinic
Other Study IDs: 10-001282
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Sleep Disordered Breathing; Cardiovascular Disease
MeSH Terms: conditions — Sleep Apnea Syndromes; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma.
Oversight: Data Monitoring Committee: No

SUMMARY:
Endothelial dysfunction, or abnormal functioning of the lining of blood vessels, appears to be a key process in the development of cardiovascular disease. Endothelial dysfunction appears to be caused by both sleep disordered breathing and obesity. As endothelial dysfunction is among the first clinical marker that predicts future cardiovascular events, understanding molecular mechanisms leading to impairment of endothelial function is very important. Endothelial function requires the proper functioning of endothelial nitric oxide synthase (eNOS). eNOS activity is tightly regulated by caveolin-1, a protein important in the formation of cellular structures called caveolae. Low levels of caveolin-1 facilitate optimal nitric oxide synthesis in endothelial cells as caveolin-1 helps to spatially organize eNOS in close proximity to signaling proteins that are important for eNOS activation. In certain diseases however, the balance of caveolin-1 and eNOS can be disrupted resulting in impaired nitric oxide synthesis and leading to endothelial dysfunction.

The investigators therefore seek to characterize levels of caveolin-1, and correlate this with the presence or absence of sleep disordered breathing, obesity, and cardiovascular disease. The current IRB protocol covers the performance of fat biopsies on subjects who have recently completed a sleep study either in the Center for Sleep Medicine or in our sleep laboratory and were found to have sleep disordered breathing or no sleep disordered breathing, subject with sleep disordered breathing who have been treated successfully with continuous positive airway pressure for 3-6 months, and subjects undergoing other studies in our lab who are obese or non-obese and subjects who have known cardiovascular disease and subjects without known cardiovascular disease.

ELIGIBILITY:
Lac of contraindication for fat biopsy, inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: With sleep disordered breathing, Without sleep disordered breathing, With cardiovascular disease, Without cardiovascular disease, Sleep disordered breathing using CPAP.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States